CLINICAL TRIAL: NCT03022188
Title: Nonfunctioning Small (≤2 cm) Neuroendocrine Pancreatic Incidentaloma: Clinical and Morphological Findings, and Therapeutic Options (IPANEMA)
Brief Title: Nonfunctioning Small (≤2 cm) Neuroendocrine Pancreatic Incidentaloma
Status: Active, not recruiting | Type: Observational
Sponsor: Société Française d'Endoscopie Digestive (Other)
Responsible Party: Principal Investigator, Gincul Rodica, Medical Doctor, Principal Investigator, Société Française d'Endoscopie Digestive
Other Study IDs: CAL-201557
Record Dates: First submitted 2017-01-10; First posted 2017-01-16 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2022-09

CONDITIONS: Neuroendocrine Tumors
Keywords: pancreatic incidentaloma; pancreatic neuroendocrine tumor; EUS-guided fine-needle aspiration; contrast-enhanced endoscopic ultrasound
MeSH Terms: conditions — Neuroendocrine Tumors; Adenoma, Islet Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: Observational

SUMMARY:
Neuroendocrine tumors (NETs) and carcinomas account for 10-15 % of all pancreatic incidentalomas. The management of pancreatic NETs depends on tumor stage and on presence or not of hormonal syndrome. The therapeutic approach for hormonally functional tumor, or large tumor (> 2 cm) with local, vascular or lymph nodes invasion, highly suggestive of malignancy, or in presence of metastasis, is well admitted: surgery is indicated or should be discussed. However, the attitude is less consensual for small (≤ 2 cm) non-functioning (NF) and non-metastatic lesions. In English, American or French recommendations, systematic surgical resection with lymphadenectomy is currently recommended in all medically fit patients. The follow-up (FU) is possible for tumors <2 cm (T1) located in the pancreatic head and for which enucleation is not feasible. Several recently published retrospective studies discuss the "non- surgical" management of the small NF incidentally detected pancreatic NETs (IPNETs) and highlight the necessity of developing guidelines for management of these patients. A strict correlation between tumor size and malignancy of these tumors was demonstrated in the single-center retrospective Italian study of Bettini and col., which included all patients with NF PNETs who underwent curative (R0) resection during 18 years. In the group of 51 patients with small size of T (2 cm or less), incidentally discovered, the majority of lesion was benign, and the authors concluded that follow-up can be proposed in patients with incidentally discovered NF PNETs ≤ 2 cm. However in despite of small size and asymptomatic character of the tumor, the rate of malignancy of NF IPNETs ≤ 2 cm was estimated to be 24 % (in 18% and 6% of cases, uncertain behaviour and carcinoma were present). Given the inherent morbidities associated with pancreatic surgery, a risk-benefit calculation may favour surveillance rather than surgery in highly selected patients. Thus, a better understanding of NF IPNETs and identification of their prognostic factors can be of help to select a subgroup of patients who could benefit from a long-term surveillance rather than a systematic surgical resection. Clearly, large prospective trials are needed to validate this approach.

DETAILED DESCRIPTION:
With increasing use of high-resolution conventional imaging, pancreatic incidentalomas are being diagnosed more frequently. In two recent surgical series, neuroendocrine tumors (NETs) and carcinomas account for 10-15 % of all pancreatic incidentalomas, the majority ( 75-90 % of cases) well differentiated. The factors affecting the behaviour of pancreatic NETs are differentiation, histological grade, staging, size and intratumoral microvascular density. In updated World Health Organization (WHO) classification, the grading system is based on tumor differentiation, the rate of proliferation and Ki-67 index. The management of pancreatic NETs depends on tumor stage and on presence or not of hormonal syndrome. By definition, the incidentally discovered pancreatic NETs (PNETs) are unassociated with hormonal syndromes (nonfunctioning) and detected in patients who undergo diagnostic evaluations for unrelated conditions.

The therapeutic approach for hormonally functional tumor, or large tumor (> 2 cm) with local, vascular or lymph nodes invasion, highly suggestive of malignancy, or in presence of metastasis, is well admitted: surgery is indicated or should be discussed.

However, the attitude is less consensual for small (≤ 2 cm) non-functioning (NF) and non-metastatic lesions. There is a paucity of literature reporting pancreatic neuroendocrine incidentalomas and their characteristics. However, given their increased incidence, they are an emerging problem and require changes in treatment guidelines. In English, American or French recommendations, systematic surgical resection with lymphadenectomy is currently recommended in all medically fit patients. The follow-up (FU) is possible for tumors <2 cm (T1) located in the pancreatic head and for which enucleation is not feasible. This therapeutic approach has two limitations: 1) the significant incidence of these tumors, because of the widespread use of routine imaging, and the improved technology of multi detector CT scan, the fortuitous discovery of small pancreatic incidentalomas is becoming more common. 2) Pancreatic surgery carries significant postoperative morbidity even in high-volume tertiary centers and even in parenchyma-preserving resection. This may results in many pancreatic resections for tumors with unknown natural history. On the other hand, the follow-up may be a factor of considerable anxiety, and carries the risk, actually difficult to assess, to let the tumor grow between two monitoring controls, with the possible evolution to the irreversible metastatic stage of the disease.

As a result, the investigators are unceasingly facing a dilemma: how to manage asymptomatic patients with small incidentally detected, potentially benign NETs? Several recently published retrospective studies discuss the "non- surgical" management of the small NF incidentally detected pancreatic NETs (IPNETs) and highlight the necessity of developing guidelines for management of these patients. A strict correlation between tumor size and malignancy of these tumors was demonstrated in the single-center retrospective Italian study of Bettini and col. , which included all patients with NF PNETs who underwent curative (R0) resection during 18 years. In the group of 51 patients with small size of T (2 cm or less), incidentally discovered, the majority of lesion was benign, and the authors concluded that follow-up can be proposed in patients with incidentally discovered NF PNETs ≤ 2 cm. However in despite of small size and asymptomatic character of the tumor, the rate of malignancy of NF IPNETs ≤ 2 cm was estimated to be 24 % (in 18% and 6% of cases, uncertain behaviour and carcinoma were present).

Given the inherent morbidities associated with pancreatic surgery, a risk-benefit calculation may favour surveillance rather than surgery in highly selected patients. Thus, a better understanding of NF IPNETs and identification of their prognostic factors can be of help to select a subgroup of patients who could benefit from a long-term surveillance rather than a systematic surgical resection. Clearly, large prospective trials are needed to validate this approach.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years old
* with a small size ≤ 2 cm (stage I) non-functioning pancreatic neuroendocrine incidentaloma, cytologically and/or histologically proved or, in case of impossibility to obtain a cyto-histological specimen, with highly suggested diagnosis by imaging (early, homogenous enhancement at computerized tomography (CT- scan) and/or magnetic resonance Imaging (MR)I and positivity at somatostatin receptor scintigraphy (SRS))
* patient ASA 1-2 (assessed according to ASA physical status classification system of American Society of Anesthesiology)
* after geriatric evaluation for the patients older than 75 y.o
* affiliated to a social security system
* with signed consent for study enrolment.

Exclusion Criteria:

* Patients < 18 years old
* Patients with NET with size > 2 cm ( stage II-IV) or NEC and/or with presence of signs suspicious of malignancy
* Patients with a functioning NET or NEC (clinical syndrome caused by excess hormonal secretion, as insulinoma or Zollinger -Ellison syndrome)
* Patients with multiple pancreatic neuroendocrine tumors
* Patients with multiple endocrine neoplasia type 1 (MEN1)
* Patients with suspicion of non- neuroendocrine tumor
* Patient ASA 3-4 (assessed according to ASA physical status classification system of American Society of Anesthesiology)
* Patients with other malignant disease under treatment or with under 5 years remission, except in situ or intramucosal carcinoma.
* Pregnant or breastfeeding women
* Patients judged not able to perform the monitoring
* Absence of signed consent for study enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with pancreatic tumors <2cm (stage 1 discovered incidentally.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-01-10 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
rate of malignancy among nonfunctioning (NF) small (≤ 2 cm) pancreatic neuroendocrine incidentalomas (PNEI). | 36 months
  * any G3 tumor *
  * G2 * or G1 * tumor with lymph node metastases and / or distant metastasis
  * G2 or G1 tumor with recurrence during the clinical and morphological surveillance after surgical treatment

SECONDARY OUTCOMES:
progression rate among NF-PNEI ≤ 2cm in case of non-surgical management | 36 months
  - significant increase of tumor size within one year > 20% on radiological examination or > 2 mm at endoscopic ultrasound ; - appearance of metastatic lymph nodes and / or distant metastases
determination of Ki67 value | 36 months
  determination of Ki67 value on cytological samples obtained by endoscopic ultrasound-guided fine-needle aspiration (EUS-FNA) and on surgical specimen
performance of contrast harmonic endoscopic ultrasound (CH-EUS) for the diagnosis of malignancy | 36 months
  assessment of sensibility (Se), specificity (Spe), positive predictive value (PPV), negative predctive value (NPV) and accuracy of CH-EUS for the diagnosis of malignancy, appreciated by tumor microvascularisation assessment during CH-EUS procédures and correlation with tumor microvascular density appreciated on surgical specimen
rate of surgical treatment, delay from diagnosis to surgery and rationale | 36 months
  number of patients having undergone surgical treatment / total number of patients included in the study ; - number of days between diagnosis and surgical treatment ,
the rate of non-surgical management and the reasons that determined the choice of this therapeutic option | 36 months
  - number of patients with non- surgical management (monitoring) / total number of patients included in the study
to assess the morbidity among the patients with surgical treatment | 36 months
  -Morbidity defined as all complication occurring after surgical resection until discharge and/or readmission, and will be grade according to the Clavien-Dindo classification. Postoperative pancreatic fistula, haemorrhage, and delayed gastric emptying were defined according to the International Study Group of Pancreatic Surgery
to assess the mortality among the patients with surgical treatment | 36 monts
  Perioperative mortality is death in relation to surgery, defined as death after surgical resection until discharge and/or readmission
to assess the overall survival (OS) among the patients with surgical treatment | 36 months
  OS defined as the time from diagnosis to death of any cause
disease specific survival (DSS) among the patients with surgical treatment | 36 months
  DSS defined as the time from diagnosis to disease-related death and censored at the last follow-up date if no events had occurred.
to assess the progression-free survival (PFS) among the patients with surgical treatment | 36 months
  PFS is the period during and after treatment in which a participant is living with a disease that does not get worse defined and is defined as the time from diagnosis until 1) loco-regional or systemic recurrence, 2) second malignancy, or 3) death from any cause; late deaths not related to cancer or its treatment are excluded
to assess the morbidity among the patients with non-surgical treatment | 36 months
  morbidity defined as all complication occurred after endoscopic ultrasound procedures until discharge and/or readmission
to assess the mortality among the patients with non-surgical treatment | 36 months
  mortality defined as death in relation to endoscopic ultrasound procedure, occured until discharge and/or readmission
to assess the overal survival (OS) among the patients with non-surgical treatment | 36 months
  OS defined as the time from diagnosis to death of any cause
to assess the disease free survival (DSS) among the patients with non-surgical treatment | 36 months
  DSS defined as the time from diagnosis to disease-related death and censored at the last follow-up date if no events had occurred.
to assess the progression-free survival (PFS) among the patients with non-surgical treatment | 36 months
  PFS is the period during and after treatment in which a participant is living with a disease that does not get worse defined and is defined as the time from diagnosis until 1) loco-regional or systemic recurrence, 2) second malignancy, or 3) death from any cause; late deaths not related to cancer or its treatment are excluded
Quality of life assessment at baseline, 12, 24 and 36 months | baseline, 12, 24 and 36 months
  The quality of life will be assessed using the 12-item Short-Form Health Survey (SF12) self- questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Rodica Gincul, MD, Principal Investigator — Société Française d'Endoscopie Digestive
Locations (22):
- Clinique Universitaire Saint Luc, Leuven, Belgium
- France (21):
  - Hopital Sud, Amiens
  - CHU Angers, Angers
  - CHRU Jean Minjoz, Besançon
  - Hopital du Haut Leveque, Bordeaux
  - Hopital Beaujon, Clichy
  - Hopital Bocage central, Dijon
  - Centre Hospitalier Lyon Sud, Lyon
  - Hopital Edouard Herriot, Lyon
  - Hopital Privé Jean Mermoz, Lyon
  - Hopital de la Timone, Marseille
  - Hopital Nord, Marseille
  - Hopital Privé Européen, Marseille
  - Hopital Saint Joseph, Marseille
  - Institut Paoli Calmette, Marseille
  - Hotel Dieu, Nantes
  - Hopital de l'archet 2, Nice
  - Clinique du Trocadero, Paris
  - Hopital Cochin, Paris
  - Hopital Européen George Pompidou, Paris
  - Hopital Robert Debré, Reims
  - CHU Rangueil, Toulouse

IPD SHARING:
Plan to Share IPD: No